CLINICAL TRIAL: NCT06516601
Title: Fulminant Cases Among Severe Community-acquired Pneumonia - an Observational Retrospective Study
Brief Title: Fulminant Severe CAP - an Observational Study
Acronym: FULMISCAP
Status: Recruiting | Type: Observational
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Confalonieri Marco, MD, Prof., University of Trieste
Other Study IDs: CEUR-2024-OS-6
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Community-acquired Pneumonia; Severe Pneumonia; ARDS, Human; Sepsis
Keywords: fulminant pneumonia; community acquired pneumonia; ARDS; sepsis; corticosteroids
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Respiratory Distress Syndrome; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — observational study, the patients received corticosteroids according to the physician on duty

SUMMARY:
Severe community-acquired pneumonia (CAP) represents a major cause of hospital mortality. Among severe CAP cases, some exhibit a rapidly progressive evolution, leading to severe ARDS/acute respiratory failure and septic shock within hours to a few days. This type of pneumonia, known as "fulminant pneumonia," is characterized by its rapid onset and deterioration, often necessitating immediate medical intervention. Despite its severity, the true incidence and optimal treatment for fulminant pneumonia are not well understood. This knowledge gap is due to the lack of attention towards pneumonia as a potential time-dependent illness and the separation of overlapping clinical topics: severe pneumonia, ARDS, and sepsis.

In clinical practice, pneumonia is the most frequent cause of both ARDS and sepsis. However, these conditions are often considered separately, combining ARDS and sepsis from various extra-pulmonary causes with those originating from pneumonia. The COVID-19 pandemic, with its vast number of severe CAP cases in a short period, has highlighted the existence of fulminant pneumonias, underscoring the need for further investigation. Recent randomized clinical trials (RCTs) and experiences from COVID-19 have suggested that early and prolonged corticosteroid administration can reduce mortality in patients with severe SARS-CoV-2 infection and severe CAP/ARDS of bacterial origin.

The aim of this observational study is to analyze the rate of fulminant pneumonia and assess the impact of early corticosteroid treatment in a multicentric population of hospitalized patients with severe pneumonia.

DETAILED DESCRIPTION:
A list of consecutive patients with severe CAP from the 5 participating centers from January 2018 to July 2024. Patients recruited for concomitant randomized clinical trials were allowed. Each Center used an early antibiotic policy (<6 hours) in case of sepsis and/or severe pneumonia diagnosis. The use of corticosteroids varied from several reasons (e.g. RCT protocol, internal policy, physician on duty with not restriction to this.

Both COVID and non-COVID patients were recruited if PaO2:FiO2 <300, bilateral community acquired pneumonia, and 2 or more of the following: increased CRP > 99mg/L, respiratory rate>25bpm or signs of respiratory distress, need for respiratory support (CPAP, MV, HFNC), creatinine>1,49mg/dl, ALT>70. Hospital-acquired and Healthcare-acquired pneumonia were excluded. Also, chronic end-stage illness (e..g. metastatic cancers, advanced neuromuscolar disorders, etc) were excluded.

The following patient caractheristics and clinical data were collected at admission: oxygenation state, vital signs, age, type of unit at admission, admission to ICU, length of hospital stay, type and duration of mechanical ventilation (MV), initial and maximal PEEP administered, ALT, WBC, platelets, Haemoglobin, presence of obesity, comorbidities, risk factors (smoking, abuse).

ELIGIBILITY:
Inclusion Criteria: severe community acquired pneumonia according to ATS/IDSA -

Exclusion Criteria: incomplete outcome data

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive patients hospitalized for severe CAP in 4 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1460 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 2days, 7days, 30days, 60days
  mortality in hospital

CONTACTS AND LOCATIONS:
Overall Officials: MARCO CONFALONIERI, MD, Principal Investigator — University of Trieste
Locations (2):
- Italy (2):
  - Marco Confalonieri, Trieste, TS
  - SC Pneumologia, Azienda Sanitaria Universitaria Giuliano-Isontina, Trieste